CLINICAL TRIAL: NCT04131647
Title: Promotion of Successful Weight Management in Overweight and Obese Veterans
Brief Title: Promotion of Weight Management
Acronym: POWER-VET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency); South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDA-013-19S
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Overweight
Keywords: Exercise; Diet; Obesity
MeSH Terms: conditions — Overweight; Motor Activity; Obesity | interventions — Body Weight Maintenance

STUDY DESIGN:
Intervention Model Description: Weight management program
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight Maintenance (Active Comparator): Heart Healthy nutrition, walking, resistance band exercise
  Interventions: Other: Weight Maintenance
- Weight Maintenance + Intermittent Fasting (Experimental): Heart Healthy nutrition, walking, resistance band exercise and intermittent fasting (2 small meals per day) one day per week for 24 weeks.
  Interventions: Other: Weight Maintenance + Intermittent Fasting

INTERVENTIONS:
Other: Weight Maintenance — Following a 12-week weight loss and exercise program, subjects will participate in a weight maintenance program of Heart Healthy nutrition, walking, and resistance band exercise
  Arms: Weight Maintenance
Other: Weight Maintenance + Intermittent Fasting — Following a 12-week weight loss and exercise program, subjects will participate in a weight maintenance program of Heart Healthy nutrition, walking, resistance band exercise and intermittent fasting (2 small meals per day) one day per week for 24 weeks.
  Arms: Weight Maintenance + Intermittent Fasting

SUMMARY:
The identification of intermittent fasting as an alternative method to traditional weight maintenance protocols could have a significant impact on preventing body weight regain common after successful weight loss, and potentially lead to a reduction in pharmaceutical and clinical costs related to the care of overweight and obese adults.

DETAILED DESCRIPTION:
The research will examine the impact of intermittent fasting to promote long term body weight maintenance following successful weight loss in overweight and obese Veterans. This research is especially relevant to the majority of Veterans who struggle with obesity and maintaining weight loss. Obesity increases the risk for storing excess calories in ectopic depots, including skeletal muscle. Intramuscular fat is related to altered substrate utilization (metabolic inflexibility) and defects in insulin sensitivity, ultimately leading to type 2 diabetes mellitus and cardiovascular disease. The objective of this proposal is to test in a randomized clinical trial the effectiveness of an intensive weight management program with and without intermittent fasting (IF) to combat weight regain and the obesity crisis in our Veterans. Further, this application proposes to examine the role of several enzymes involved in skeletal muscle fatty acid oxidation as a mechanism for efficacious long term weight management.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* 50-75 years of age
* BMI: 25-40 kg/m2
* Postmenopausal status for women

Exclusion Criteria:

* Uncontrolled diabetes (HbA1c >10% or the current use of insulin)
* Neurologic, musculoskeletal, or other condition that limits subject's ability to complete study physical assessments
* Active inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignant, and psychiatric disease
* Weight change within the past month of >5 kg
* Self-reported alcohol or drug abuse
* Anti-coagulant medication for muscle biopsies only Impaired renal function (creatinine > 1.5 mg/dl) History or evidence of serious liver disease (LFTs > 2.5 x WNL)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, after 12 weeks of weight loss+exercise, at 36-week weight maintenance, and 48-week follow-up
  weight in kg

SECONDARY OUTCOMES:
Change in Gait Speed | Baseline, after 12 weeks of weight loss+exercise, at 36-week weight maintenance, and 48-week follow-up
  Fastest comfortable walking speed over 4 meters. Units are m/sec
Change in body fat | Baseline, after 12 weeks of weight loss+exercise, and at 36-week weight maintenance
  abdominal fat area, in cm2
Change in LPL | Baseline, after 12 weeks of weight loss+exercise, and at 36-week weight maintenance
  skeletal muscle lipoprotein lipase in nmol/min/ mg protein

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04131647/ICF_000.pdf